CLINICAL TRIAL: NCT05084404
Title: Phase II Physician-initiated Clinical Trial Investigating the Efficacy and Safety of Guanabenz Acetate for Non-alcoholic Fatty Liver Disease Associated With Hypertension
Brief Title: Efficacy and Safety of Guanabenz for Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yokohama City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YCU-21001
Record Dates: First submitted 2021-09-24; First posted 2021-10-19 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Guanabenz; Phase 2 trial
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Guanabenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 mg/day of WY-8678 (guanabenz acetate) (Experimental)
  Interventions: Drug: Experimental: 4 mg/day of WY-8678 (guanabenz acetate)
- 8 mg/day of WY-8678 (guanabenz acetate) (Experimental)
  Interventions: Drug: Experimental: 8 mg/day of WY-8678 (guanabenz acetate)

INTERVENTIONS:
Drug: Experimental: 4 mg/day of WY-8678 (guanabenz acetate) — Patients with nonalcoholic fatty liver disease are administered 4 mg/day of WY-8678 (guanabenz acetate) twice daily for 16 weeks
  Arms: 4 mg/day of WY-8678 (guanabenz acetate)
Drug: Experimental: 8 mg/day of WY-8678 (guanabenz acetate) — Patients with nonalcoholic fatty liver disease are administered 8 mg/day of WY-8678 (guanabenz acetate) twice daily for 16 weeks
  Arms: 8 mg/day of WY-8678 (guanabenz acetate)

SUMMARY:
To investigate the efficacy and safety of 4 mg/day of WY-8678 (guanabenz acetate) and 8 mg/day of WY-8678 (guanabenz acetate) in patients with non-alcoholic fatty liver disease/non-alcoholic steatohepatitis (NAFLD/NASH patients) with hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have received a full explanation about this study and who have provided written consent.
2. Patients ≥ 20 years of age ≤ 75 years of age at the time consent was provided.
3. Patients diagnosed with essential hypertension and whose systolic blood pressure at the time of screening is ≥ 130 mmHg and/or diastolic blood pressure is ≥ 85 mmHg (according to the diagnostic criteria for metabolic syndrome)
4. Patients diagnosed with NAFLD/NASH who meet the following criteria (1) or (2) (1) Patients diagnosed with NAFLD who meet the following three criteria: ・Diagnostic imaging or histological evidence of fatty liver, ・Alcohol intake < 30 g/day for men and < 20 g/day for women for 12 or more consecutive weeks one year before screening, ・Absence of other factors that cause fattening or chronic liver disease. (2) Patients with a definitive diagnosis of NASH by biopsy within 32 weeks before screening * The definitive diagnostic criteria for NASH are defined as a fibrosis stage in liver biopsy in the evaluation using the "NASH Clinical Research Network (CRN) criteria" by an F1-F3 pathologist and a NAFLD activity score (NAS) ≥4 points (each item has one or more points): ・Steatosis (0-3 points)

   * Ballooning (0-2 points)
   * Inflammation in the lobules (0-3 points)
5. Patients with magnetic resonance imaging (MRI)-proton density fat fraction (PDFF) liver fat mass ≥ 8% at screening.
6. Patients with magnetic resonance elastography (MRE) value ≤ 3.6 kPa at screening.
7. Patients with a body mass index (BMI) ≥ 25 kg/m2 at the time of screening.
8. Patients receiving diet or exercise therapy 12 weeks before screening, with no improvement.
9. Patients who are willing to maintain a stable diet and physical activity during the clinical trial.

Exclusion Criteria:

1. Pregnant, lactating, potentially pregnant women, or patients who do not agree to contraception during the trial period.
2. Patients who have taken guanabenz acetate within 16 weeks prior to screening or who have participated in other clinical studies (observational studies are excluded).

3. Patients with drug allergies to guanabenz acetate. 4. Patients with liver failure or cirrhosis. 5. Patients with the following laboratory test values:

(1) Alanine aminotransferase (ALT) > 430 IU/L (males) or > 240 IU/L (female); or aspartate aminotransferase (AST) > 300 IU/L (males and females) (2) Prothrombin time-international normalized ratio (PT-INR) ≥ 1.5 (excluding anticoagulant therapy) (3) Total bilirubin value > 2.0 mg/dL (excluding definitive diagnosis of Gilbert syndrome) (4) Platelet count < 80,000/μL (5) Estimated glomerular filtration ratio (eGFR) < 45 (calculated by body surface area correction: standardized eGFR) 6. Patients with a history of acute or chronic liver disease other than NAFLD/NASH and complications:

1. Patients suffering from hepatitis B (defined by hepatitis B surface (HBs) antigen positive at the time of screening) or hepatitis C (defined by hepatitis C virus (HCV) antibody positive at the time of screening). However, anti-HCV antibody positive patients who are judged to be negative for hepatitis C virus ribonucleic acid (HCV-RNA) can be registered if they can be confirmed to be negative for at least one year before screening.
2. Patients with autoimmune hepatitis.
3. Patients with primary biliary cholangitis, primary sclerosing cholangitis, Wilson's disease, α1-antitrypsin deficiency, hemochromatosis or iron overload, drug-induced or alcoholic liver disease, or a history of known biliary atresia.
4. Patients with suspicion or definitive diagnosis of hepatocellular carcinoma. 7. Patients with a history of human immunodeficiency virus (HIV) infection. 8. Patients with findings of portal hypertension (complications: ascites, hepatic encephalopathy, varicose veins, splenomegaly).

9. Patients with a history of NAFLD-related drugs (amiodarone, methotrexate, systemic glucocorticoids, tetracycline, tamoxifen, higher doses of estrogen, anabolic steroids or valproic acid than used for hormone replacement) or other hepatotoxins for at least 4 weeks prior to screening.

10. Patients who have used the following drugs:

1. Patients who used insulin, glucagon-like peptide-1 (GLP-1) receptor agonists, SGLT2 inhibitors, or thiazolidine 12 weeks before screening,
2. Patients who used ursodeoxycholic acid or vitamin E 12 weeks before screening,
3. Patients whose doses of dyslipidemia drugs or antihypertensive drugs were changed 12 weeks before screening,
4. Patients whose dose of oral diabetes treatment drug (dipeptidyl peptidase 4 [DPP-4] inhibitor, sulfonylurea [SU] preparation, α-glucosidase inhibitor, metformin) was changed 12 weeks before screening,
5. Patients who used drugs known to have a significant effect on body weight (including over-the-counter drugs for weight loss) 12 weeks before screening,
6. Patients using central nervous system depressants (barbital, sodium thiopental, morphine hydrochloride hydrate, brotizolam, diazepam, etc.).

11. Patients with 10% weight change 24 weeks before screening. 12. Patients scheduled to undergo surgery after obesity surgery (such as gastroplasty and Roux-en-Y gastric bypass surgery) or during the trial period.

13. Patients with a history of type 1 diabetes. 14. Patients with hemoglobin A1c (HbA1c) > 9.5% at screening or with uncontrolled type 2 diabetes.

15. Patients with hyperthyroidism or hypothyroidism, or screening results showing thyroid dysfunction. However, for hypothyroidism, registration is possible if thyroid replacement therapy is received 12 weeks before screening and the test values are stable.

16. Patients with a history of New York heart association functional classification (NYHA classification) class III or IV heart failure due to factors other than hypertension.

17. Patients with a history of myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting, or stroke or major surgery 24 weeks before screening.

18. Patients with a history of substance abuse. 19. Patients with malignant tumors. However, patients who have undergone radical surgery, patients who have completed chemotherapy/radiation therapy, and patients who are undergoing hormone therapy can be registered.

20. Patients with known intolerance to MRI or patients who are contraindicated for MRI examination.

21. Other patients who the principal investigator or sub-investigator deems inappropriate for conducting this clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of those where the liver fat content (%) measured by MRI-PDFF at 16 weeks decreased by ≥ 3.46% from baseline (%) | Week 16
  MRI-PDFF

SECONDARY OUTCOMES:
Percentage of those where the liver fat content (%) measured by MRI-PDFF at 16 weeks decreased by 3.46% or more from baseline for 4 mg group and 8 mg group (%) | Week 16
  MRI-PDFF
The absolute change in liver fat content measured by MRI-PDFF | Week 16
  MRI-PDFF
Rate of change in ALT | Week 16
  Serum
Rate of change in AST | Week 16
  Serum
Rate of change in gamma-glutamyl transferase (γ-GTP) | Week 16
  Serum
Rate of change in weight | Week 16
  Body weight
Rate of change in blood lipids | Week 16
  Serum. Blood lipids defined as (chylomicron cholesterol, chylomicron triglyceride, lipoprotein cholesterol, low-density lipoprotein [LDL] triglyceride, very low-density lipoprotein [VLDL] cholesterol, VLDL triglyceride, free cholesterol, apoprotein A1, apoprotein B, adipsin, free fatty acid).
Rate of change in insulin resistance (HOMA-IR) | Week 16
  Blood
Rate of change in liver stiffness | Week 16
  MR elastography
Rate of change in fibrosis markers (enhanced liver fibrosis [ELF] score) | Week 16
  Serum
Rate of change in fibrosis markers (enhanced liver fibrosis Fibrosis-4 [FIB-4]) | Week 16
  Serum
Occurrence rate of adverse events | Week 0-16
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Yokohama City University, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwaki M, Kessoku T, Tanaka K, Ozaki A, Kasai Y, Yamamoto A, Takahashi K, Kobayashi T, Nogami A, Honda Y, Ogawa Y, Imajo K, Yoneda M, Kobayashi N, Saito S, Nakajima A. Efficacy and safety of guanabenz acetate treatment for non-alcoholic fatty liver disease: a study protocol for a randomised investigator-initiated phase IIa study. BMJ Open. 2022 Jul 12;12(7):e060335. doi: 10.1136/bmjopen-2021-060335. PMID 35820743